CLINICAL TRIAL: NCT00870727
Title: Pharmacotherapy of Pervasive Developmental Disorders
Brief Title: Study of Aripiprazole in the Treatment of Pervasive Developmental Disorders
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0805-26; MH 082119
Record Dates: First submitted 2009-02-02; First posted 2009-03-27 (Estimated); Results first posted 2018-11-28 (Actual); Last update posted 2019-01-02 (Actual); Status verified 2018-03

CONDITIONS: Pervasive Developmental Disorder
Keywords: PDD NOS
MeSH Terms: conditions — Child Development Disorders, Pervasive | interventions — Aripiprazole; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1. Aripiprazole oral product (Experimental): Participants will receive Aripiprazole oral product with a minimum dose of 2 mg per day to a maximum dose of 20 mg per day over 8-weeks of treatment.
  Interventions: Drug: Aripiprazole oral product
- Arm 2. Placebo oral capsule (Placebo Comparator): Participants will receive matching (identical in size and appearance to study drug) placebo oral capsules over 8-weeks of treatment.
  Interventions: Drug: Placebo oral capsule

INTERVENTIONS:
Drug: Aripiprazole oral product — Minimum dose of 2 mg per day to a maximum dose of 20 mg per day over 8-weeks of treatment.
  Other Names: Abilify
  Arms: Arm 1. Aripiprazole oral product
Drug: Placebo oral capsule — Placebo will be identical in size and appearance to study drug.
  Other Names: Sugar pill
  Arms: Arm 2. Placebo oral capsule

SUMMARY:
The purpose of this study is to develop a better tolerated and more effective pharmacologic treatment with individuals with Pervasive Developmental Disorder. This is a double-blind, placebo-controlled study of aripiprazole in the management of the maladaptive behaviors of Pervasive Developmental Disorder. The investigators hypothesize that aripiprazole will be more effective than placebo for reducing aggression, tantrum and self-injurious behavior in children with Pervasive Developmental Disorder.

DETAILED DESCRIPTION:
Pervasive developmental disorders (PDDs) are characterized by severe impairments in social interaction and communication in addition to restricted patterns of interests and activities. Research suggests that a dysregulation of the dopamine and serotonin systems contributes to these interfering behaviors in individuals with PDD. After benefits of typical neuroleptics were reported in subjects with PDD, research shifted to the atypical antipsychotics which have been shown to be better tolerated and effective in this population. However, the atypical antipsychotics have also been associated with adverse effects. Thus there remains a need for a novel pharmacotherapy that would be safe and effective for children and adolescents with PDDs. The primary objectives of this study are to determine whether aripiprazole is effective and well tolerated for irritability in children and adolescents with PDD not otherwise specified (NOS) during an 8-week acute phase and whether the effectiveness and tolerability of aripiprazole is maintained during a 16-week continuation phase.

ELIGIBILITY:
Inclusion Criteria:

* Male and female outpatients between the ages of 5 and 17 years and greater than or equal to 15 kg body weight.
* Diagnostic and Statistical Manual of Mental Disorders Fourth Edition, Text Revised (DSM-IV-TR) diagnosis of Pervasive Developmental Disorder Not Otherwise Specified (PDD NOS).
* Psychotropic medication-free for at least 2 days prior to screening laboratory tests and electrocardiogram (ECG).
* Significant irritability as determined by a Clinical Global Impression Severity score of greater or equal to 4 (Moderately ill) and a score of equal to or greater than 18 on the Aberrant Behavior Checklist Irritability Subscale.
* Intelligence quotient (IQ) of equal to or greater than 50 based on the Wechsler Intelligence Scale for Children (WISC), 4th edition; the Leiter International Test of Intelligence-Revised will be used if a child is nonverbal but thought to have an IQ greater than or equal to 50.

Exclusion Criteria:

* DSM-IV-TR diagnosis other than PDD NOS (autistic disorder, Asperger's disorder, Rett's disorder, or childhood disintegrative disorder), schizophrenia, bipolar disorder or substance abuse within the last 6 months.
* Comorbid disorder with possible association to autism (e.g., Fragile X Syndrome, Tuberous Sclerosis).
* A significant medical condition such as heart, liver, renal, or pulmonary disease, or a seizure disorder, as determined by history, physical examination, or laboratory testing.
* Subjects with an active seizure disorder (history of febrile seizures in early childhood will be considered.
* Females with a positive urine pregnancy test.
* Evidence of a prior adequate trial of aripiprazole (defined as equal to or greater than 2 weeks at equal to or greater than 5 mg per day. When there is not evidence of a prior adequate trial, subjects must be medication-free for a least 2 weeks prior to baseline.
* History of neuroleptic malignant syndrome.
* Subjects who, in the opinion of the investigator, are unsuitable in any other way to participate in this study, including being unable to comply with the requirements of the study for any reason.
* Hypersensitivity to aripiprazole [e.g., allergic response or serious adverse effect] (significant tachycardia).

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 33 (Actual)
Dates: Start 2009-02; Primary Completion 2015-03 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly A. Stigler, MD, Principal Investigator — Indiana University
Locations (1):
- Riley Hospital for Children, Christian Sarkine Autism Treatment Center, Indianapolis, Indiana, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1. Aripiprazole Oral Product: Participants will receive Aripiprazole oral product with a minimum dose of 2 mg per day to a maximum dose of 20 mg per day over 8-weeks of treatment.
  Aripiprazole oral product: Minimum dose of 2mg per day to a maximum of 20 mg per day over 8-weeks of treatment.
- Arm 2. Placebo Oral Capsule: Participants will receive matching (identical in size and appearance to study drug) placebo oral capsules over 8-weeks of treatment.
  Placebo oral capsule: Placebo will identical in size and appearance to study drug.
Period: Overall Study
Arm/Group | Arm 1. Aripiprazole Oral Product | Arm 2. Placebo Oral Capsule
Started | 17 | 16
Completed | 16 | 11
Not Completed | 1 | 5
Not completed — Lost to Follow-up | 0 | 1
Not completed — Lack of Efficacy | 1 | 3
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1. Aripiprazole Oral Product | Arm 2. Placebo Oral Capsule | Total
Number analyzed (Participants) | 17 | 16 | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.8 (3.0) | 9.5 (2.3) | 9.6 (2.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 5 | 7
  Male | 15 | 11 | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 16 | 16 | 32
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 3 | 4
  White | 15 | 11 | 26
  More than one race | 1 | 2 | 3
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 17 | 16 | 33

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Improved as Measured by the Clinical Global Impression-Global Improvement Scale (Improvement Defined as CGI-I=1 or CGI-I=2)
Description: Clinical Global Impressions (Guy, 1976) global improvement (CGI-I) is designed to take into account all factors to arrive at an assessment of response to treatment. The CGI-I scale ranges from 1 to 7, with lower scores indicating greater improvement (1=very much improved and 2=much improved). Participants with a CGI-I score of 1 or 2 were classified as improved. Four participants assigned to placebo completed an exit interview prior to week 8. One participant assigned to placebo and one participant assigned to aripiprazole withdrew from the study without completing an exit interview.
Time Frame: Double-blind phase study exit - up to 8 weeks
Population: All randomized study participants who completed an exit interview
Measure: Number; unit: participants
Arm/Group | Arm 1. Aripiprazole Oral Product | Arm 2. Placebo Oral Capsule
Number analyzed (Participants) | 16 | 15
participants | 11 | 3

2. Primary Outcome: Mean Post-baseline Aberrant Behavior Checklist Irritability Subscale Score, Parent Report, Double-blind Phase
Description: The Aberrant Behavior Checklist (ABC) is a symptom checklist for assessing problem behaviors in individuals ages 6 to 54 years-old with mental retardation. The full ABC is a 58-item parent rating with five factors: Irritability, Social Withdrawal, Stereotypy, Hyperactivity and Inappropriate Speech. It has been used as a primary outcome measure in several trials in children with developmental disabilities. The interpretation of the tool and its subscales is that a greater number of items indicates greater severity. The range of scores for the Irritability subscale is 0 to 45. Means were estimated using a repeated measures linear regression model with treatment group, baseline score, study week (in categories), and Tanner stage as covariates. A linear contrast estimated the average across study timepoints. Confidence intervals reflect a Bonferroni multiple testing correction accounting for the selection of two primary outcomes.
Time Frame: Weeks 1, 2, 3, 4, 6 and 8
Population: All randomized study participants
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Arm 1. Aripiprazole Oral Product | Arm 2. Placebo Oral Capsule
Number analyzed (Participants) | 17 | 16
units on a scale | 18.3 [14.2 to 22.5] | 26.4 [22.1 to 30.8]

3. Secondary Outcome: Mean Post-baseline Aberrant Behavior Checklist Hyperactivity Subscale Score, Parent Report, Double-blind Phase
Description: The Aberrant Behavior Checklist (ABC) is a symptom checklist for assessing problem behaviors in individuals ages 6 to 54 years-old with mental retardation. The full ABC is a 58-item parent rating with five factors: Irritability, Social Withdrawal, Stereotypy, Hyperactivity and Inappropriate Speech. The 16-item Hyperactivity subscale covers overactivity (7 items), impulsiveness (2 items), inattention (3 items) and noncompliance (4 items). It has been used as a primary outcome measure in several trials in children with developmental disabilities. The interpretation of the tool and its subscales is that a greater number of items indicates greater severity. The range of scores is 0 to 48 on the Hyperactivity subscale. Means were estimated using a repeated measures linear regression model with treatment group, baseline score, study week (in categories), and Tanner stage as covariates. A linear contrast estimated the average across study timepoints.
Time Frame: Weeks 1, 2, 3, 4, 6 and 8
Population: All randomized study participants
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Arm 1. Aripiprazole Oral Product | Arm 2. Placebo Oral Capsule
Number analyzed (Participants) | 17 | 16
units on a scale | 23.8 [19.7 to 28.0] | 29.4 [25.2 to 33.8]

4. Secondary Outcome: Mean Post-baseline Aberrant Behavior Checklist Inappropriate Speech Subscale Score, Parent Report, Double-blind Phase
Description: The Aberrant Behavior Checklist (ABC) is a symptom checklist for assessing problem behaviors in individuals ages 6 to 54 years-old with mental retardation. The full ABC is a 58-item parent rating with five factors: Irritability, Social Withdrawal, Stereotypy, Hyperactivity and Inappropriate Speech. It has been used as a primary outcome measure in several trials in children with developmental disabilities. The interpretation of the tool and its subscales is that a greater number of items indicates greater severity. The range of scores for the Inappropriate Speech subscale is 0 to 12. Means were estimated using a repeated measures linear regression model with treatment group, baseline score, study week (in categories), and Tanner stage as covariates. A linear contrast estimated the average across study timepoints.
Time Frame: Weeks 1, 2, 3, 4, 6 and 8
Population: All randomized study participants
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Arm 1. Aripiprazole Oral Product | Arm 2. Placebo Oral Capsule
Number analyzed (Participants) | 17 | 16
units on a scale | 4.6 [3.8 to 5.4] | 6.0 [5.2 to 6.8]

5. Secondary Outcome: Mean Post-baseline Aberrant Behavior Checklist Social Withdrawal Subscale Score, Parent Report, Double-blind Phase
Description: The Aberrant Behavior Checklist (ABC) is a symptom checklist for assessing problem behaviors in individuals ages 6 to 54 years-old with mental retardation. The full ABC is a 58-item Parent rating with five factors: Irritability, Social Withdrawal, Stereotypy, Hyperactivity and Inappropriate Speech. It has been used as a primary outcome measure in several trials in children with developmental disabilities. The interpretation of the tool and its subscales is that a greater number of items indicates greater severity. The range of scores for the Social Withdrawal subscale is 0 to 48. Means were estimated using a repeated measures linear regression model with treatment group, baseline score, study week (in categories), and Tanner stage as covariates. A linear contrast estimated the average across study timepoints.
Time Frame: Weeks 1, 2, 3, 4, 6 and 8
Population: All randomized study participants
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Arm 1. Aripiprazole Oral Product | Arm 2. Placebo Oral Capsule
Number analyzed (Participants) | 17 | 16
units on a scale | 6.1 [3.4 to 8.7] | 9.6 [6.8 to 12.4]

6. Secondary Outcome: Mean Post-baseline Aberrant Behavior Checklist Stereotypy Subscale Score, Parent Report, Double-blind Phase
Description: The Aberrant Behavior Checklist (ABC) is a symptom checklist for assessing problem behaviors in individuals ages 6 to 54 years-old with mental retardation. The full ABC is a 58-item parent rating with five factors: Irritability, Social Withdrawal, Stereotypy, Hyperactivity and Inappropriate Speech. It has been used as a primary outcome measure in several trials in children with developmental disabilities. The interpretation of the tool and its subscales is that a greater number of items indicates greater severity. The range of scores for the Stereotypy subscale is 0 to 21. Means were estimated using a repeated measures linear regression model with treatment group, baseline score, study week (in categories), and Tanner stage as covariates. A linear contrast estimated the average across study timepoints.
Time Frame: Weeks 1, 2, 3, 4, 6 and 8
Population: All randomized study participants
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Arm 1. Aripiprazole Oral Product | Arm 2. Placebo Oral Capsule
Number analyzed (Participants) | 17 | 16
units on a scale | 3.9 [2.6 to 5.3] | 5.3 [3.9 to 6.7]

ADVERSE EVENTS:
Time Frame: Eight weeks or at the time of latest data collection.
Description: Adverse event information was collected via a structured side effect rating scale completed with the participant and their primary caregiver. This included a list of side-effects that have been reported with aripiprazole at a rate greater than 1%. The physician also asked about any visits to the doctor, new medication use, or any other complaints. Events that were not present at baseline and occurred or worsened after the date of randomization are reported.
Arm/Group | Arm 1. Aripiprazole Oral Product | Arm 2. Placebo Oral Capsule
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/16
Other Adverse Events (participants affected / at risk) | 16/17 | 13/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1. Aripiprazole Oral Product (N=17) | Arm 2. Placebo Oral Capsule (N=16)
Constipation (Gastrointestinal disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Stomach or abdominal discomfort (Gastrointestinal disorders) | 4 | 3
Vomiting (Gastrointestinal disorders) | 0 | 2
Appetite decrease (General disorders) | 3 | 0
Appetite increase (General disorders) | 6 | 2
Dry mouth (General disorders) | 1 | 0
Fever (General disorders) | 1 | 1
Hypersalivation (General disorders) | 4 | 0
Increased thirst (General disorders) | 0 | 1
Other Pain (General disorders) | 1 | 0
Sedation/Drowsiness (General disorders) | 3 | 1
Tiredness/Fatigue (General disorders) | 5 | 3
Allergies Not Otherwise Specified (Immune system disorders) | 0 | 1
Flu or upper respiratory problems (Infections and infestations) | 0 | 2
Nasal congestion or Cold (Infections and infestations) | 2 | 6
Sore throat (Infections and infestations) | 0 | 1
Weight gain (Metabolism and nutrition disorders) | 3 | 1
Weight loss (Metabolism and nutrition disorders) | 1 | 0
Muscle/bone/joint pain/condition (Musculoskeletal and connective tissue disorders) | 1 | 1
Headache (Nervous system disorders) | 5 | 5
Tremor (Nervous system disorders) | 0 | 1
Unspecified or not otherwise listed head (Nervous system disorders) | 1 | 0
Anxiety/Nervousness/Worry (Psychiatric disorders) | 0 | 1
Change in speech (Psychiatric disorders) | 1 | 1
Concentration difficulty (Psychiatric disorders) | 1 | 0
Daydreaming (Psychiatric disorders) | 2 | 0
Difficulty falling asleep (Psychiatric disorders) | 1 | 3
Echolalia (Psychiatric disorders) | 0 | 1
Emotional outburst (Psychiatric disorders) | 1 | 0
Hypertalkativeness (Psychiatric disorders) | 1 | 0
Increased motor activity (Psychiatric disorders) | 2 | 0
Interrupted sleep/other sleep problems (Psychiatric disorders) | 2 | 3
Irritability (Psychiatric disorders) | 0 | 5
Restlessness/Agitation including fidgety (Psychiatric disorders) | 2 | 0
Stereotypy (Psychiatric disorders) | 1 | 0
Unspecified or not otherwise listed psych (Psychiatric disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Generalized rash (Skin and subcutaneous tissue disorders) | 1 | 0
Localized rash (Skin and subcutaneous tissue disorders) | 1 | 0
Intermittent nosebleed (Vascular disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
The PI who conducted the trial left the institution, Indiana University, prior to data analysis. The institution negotiated/executed a data transfer agreement for the PI's primary mentor, Dr. Christopher McDougle, to analyze the data on her behalf.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No